CLINICAL TRIAL: NCT06788145
Title: Enhancing Social Connections Among Rural Community Members With Disordered Eating
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Principal Investigator, Caitlin Martin-Wagar, Assistant Professor, University of Montana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2024-307
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Eating Disorders (Excluding Anorexia Nervosa); Disordered Eating; Disordered Eating Behaviors; Eating Disorder Symptom
Keywords: eating disorder; disordered eating
MeSH Terms: conditions — Feeding and Eating Disorders; Disordered Eating Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Session Intervention (Experimental)
  Interventions: Behavioral: Social Support Single-Session Intervention

INTERVENTIONS:
Behavioral: Social Support Single-Session Intervention — Single-session intervention to increase self-efficacy, social support, help-seeking, and recovery-oriented behaviors to address disordered eating.

SUMMARY:
This study is about testing a short program that uses social support to help people with disordered eating. The goal is to see if this program can help people build better habits and feel better about eating while reducing harmful symptoms. In the long run, this project wants to make it easier for people with eating problems to get help and recover, especially for those in rural areas or other groups who don't often get the care they need. Participants will complete self-report measures online, and complete a digital single-session program.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years old)
* disordered eating
* live in the United States of America

Exclusion Criteria:

* BMI below 18.5

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
eating disorder symptoms | 1 month post-intervention
  As measured for the Eating Disorder Examination Questionnaire

SECONDARY OUTCOMES:
Help-seeking | 1 month post-intervention
  As measured by the General Help Seeking Questionnaire and qualitative help-seeking behavioral questions.
Self-efficacy | 1 month post-intervention
  As measured by the General Self-Efficacy scale
Social support and sense of community | 1 month post-intervention
  As measured by the MOS Social Support Survey and Sense of Community Index
Personal Growth | 1 month post-intervention
  As measured by the Personal Growth Initiative

OTHER OUTCOMES:
Program feedback | 1 month post-intervention
  As measured by the Program Feedback Scale
Acceptability | 1 month post-intervention
  As measured by the Credibility and Expectancy Questionnaire, and qualitative open-ended questions

IPD SHARING:
Plan to Share IPD: Undecided